CLINICAL TRIAL: NCT01208246
Title: Impact of Pelvic Floor Musculature on Peripartum Outcomes: A Prospective Study
Brief Title: Impact of Pelvic Floor Musculature on Peripartum Outcomes
Acronym: PregUS
Status: Completed | Type: Observational
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Tulin Ozcan MD, Associate Professor, University of Rochester
Other Study IDs: 31522
Record Dates: First submitted 2010-09-22; First posted 2010-09-23 (Estimated); Last update posted 2014-02-21 (Estimated); Status verified 2014-02

CONDITIONS: Pregnancy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to understand the effect of the pregnancy on the muscles in the pelvis. The purpose of this study is to evaluate the pelvic muscle changes related to pregnancy; to assess if the ability to squeeze and relax these muscles has any effect on delivery mode and if there are any injuries to the pelvic muscles.

DETAILED DESCRIPTION:
Healthy women who are pregnant with their first child will be included in the study. Information about their general health will be gathered. These women will be screened for pelvic disorders at the start and end of study. Three-dimensional ultrasound will be performed three times: 12-24 weeks, 34-39 weeks and 4-6 weeks after delivery. Fetal measurements will be included in the third trimester ultrasound for prediction of estimated birth weight. The relationship of the predicted fetal weight and the likelihood of having a successful vaginal delivery will be studied. Images will be analyzed for pelvic muscles function and injuries. Information regarding the length of labor, types of delivery and vaginal tears will be gathered. The information obtained will be analyzed to look for the strength of correlation of variables to the outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Primiparous or should not have given birth to a fetus older than 12 weeks.
* Singleton pregnancy.
* Age more than or equal to 18 years.
* Basal mass index between 18 - 40 kg/m2.
* Must plan to deliver at Strong Memorial Hospital at the University of Rochester Medical Center.

Exclusion Criteria:

* Basal mass index more than 40 kg/m2.
* Presence of current or prior history of cervical incompetence.
* Presence of diabetes mellitus (type I or type II).
* Presence of connective-tissue disorders such as Systemic lupus erythematosus, Rheumatoid Arthritis, or Sjogren's disease.
* Presence of neuromuscular disorders such as myasthenia gravis and neuropathies.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Prenatal visits
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2010-04; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Serial changes in pelvic floor anatomy and function | 12-24 weeks, 34-39 weeks gestation, and 4-6 weeks postpartum
  To evaluate the serial changes in pelvic floor anatomy and function during the second, third trimester of pregnancy and in the postpartum period.

CONTACTS AND LOCATIONS:
Overall Officials: Tulin Ozcan, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States